CLINICAL TRIAL: NCT05573139
Title: Reliability and Validation of New Manual Dynamometer to Measure Lower Limb Strength: Clinical Study
Brief Title: Reliability and Validation of New Manual Dynamometer to Measure Lower Limb Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MEDEOR
Record Dates: First submitted 2022-04-27; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Muscle Strength; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- muscle strength assessment (Experimental)
  Interventions: Diagnostic Test: Assessment of muscle strength by manual dynamometry

INTERVENTIONS:
Diagnostic Test: Assessment of muscle strength by manual dynamometry — The reliability and validation of a new manual dynamometer was verified, compared to one already used, in the muscle groups: knee extensors and flexors; hip extensors, flexors, abductors, adductors, internal and external rotators.

SUMMARY:
INTRODUCTION: There are several ways to assess muscle strength: not only subjective ways, but also high standard equipment, such as isokinetic dynamometers. These, however, are expensive, and require extensive training. Over the years, manual dynamometers were produced, portable equipment that simplify its use. Among them, a national equipment was developed, but its reliability and validation are yet to be confirmed, compared to equipment already used, such as the Lafayette®. OBJECTIVE: Assess the reliability of a new manual dynamometer - Medeor® device (SP Tech model) -, in relation to the gold standard, Lafayette® device (model 01165), already validated, in the evaluation of muscle strength of the knee and hip groups. METHODS: A total of 26 recruits of both sexes were selected. Muscle strength was measured by Lafayette® and Medeor® dynamometers in the following groups: knee flexors and extensors; flexors, extensors, abductors, adductors, hips internal and external rotators. Each data was collected 3 times, and then the average was calculated.

DETAILED DESCRIPTION:
Keywords: Muscle Strength; Muscle Strength Dynamometer; Lower Extremity.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 year
* both sex
* Healthy

Exclusion Criteria:

* individual who practiced physical activity,
* cognitive disability
* osteomioarticular diseases in lower limb and/or spine
* rheumatic or cardiorespiratory disease

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Muscle strength assessment by hand dynamometer of the hip | 1 day (single assessment)
  Assessment of muscle strength by hand dynamometer of the hip
Muscle strength assessment by hand dynamometer of the knee | 1 day (single assessment)
  Assessment of muscle strength by hand dynamometer of the knee

CONTACTS AND LOCATIONS:
Locations (1):
- Claudio Cazarini Júnior, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No